CLINICAL TRIAL: NCT05853783
Title: Evaluation of Oral Potentially Malignant Disorders (OPMDs) with STRATICYTE™
Status: Recruiting | Type: Observational
Sponsor: Proteocyte Diagnostics Inc. (Industry)
Collaborators: The University of Texas Health Science Center, Houston (Other); Loma Linda University (Other); Minnesota Oral & Facial Surgery (Unknown); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: PRO-STR-PPOEL-2
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Mouth Diseases
Keywords: Leukoplakia; Erythroplakia; Erythroleukoplakia; Lesion; Oral epithelial dysplasia; S100A7 biomarker; S100A7 Immunohistochemistry Signature-based; Early Diagnosis; STRATICYTE; Oral neoplasia; Oral epithelial atypia; Hyperplasia; Hyperkeratosis; Potentially premalignant oral epithelial lesion; Oral potentially malignant disorders; Mild dysplasia; Moderate dysplasia; Severe dysplasia; Low-grade dyspalsia; High-grade dysplasia; Personalized medicine; Predictive Assay; Whole slide imaging; Computational pathology; Digital pathology; Oral potentially malignant lesion
MeSH Terms: conditions — Mouth Diseases; Leukoplakia; Erythroplasia; Disease; Hyperplasia; Keratoderma, Palmoplantar, Epidermolytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — FFPE specimens immunohistochemically stained with S100A7
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OPMDs that progressed to OSCC: No dysplasia, mild, moderate, severe dysplasia, CIS
  Interventions: Other: STRATICYTE™ Test
- OPMDs that did not progress to OSCC: No dysplasia, mild, moderate, severe dysplasia, CIS
  Interventions: Other: STRATICYTE™ Test

INTERVENTIONS:
Other: STRATICYTE™ Test — Assessment for risk of progression to oral cancer
  Other Names: S100A7 Immunohistochemistry Signature-based Test

SUMMARY:
The purpose of this study is to validate the ability of the STRATICYTE™ predictive model to predict the transformation of oral potentially malignant disorders (OPMDs) to oral squamous cell carcinoma (OSCC) in a retrospective cohort of patients who received biopsies.

DETAILED DESCRIPTION:
The study objectives are to:

1. Evaluate STRATICYTE™ sensitivity and specificity in a cohort of patients that meet the inclusion/exclusion criteria.
2. Identify patient and clinical characteristics influencing the sensitivity and specificity of the STRATICYTE™ model.
3. Estimate the correlation between STRATICYTE™ outcome and time to a positive diagnosis of oral cancer.

ELIGIBILITY:
Inclusion Criteria:

* From the archive, any patient who presents with clinically evident oral lesions and biopsy-proven dysplasia (punch or scalpel biopsies; any grade or classification system)
* Patients with initial oral lesions with epithelial atypia suspicious for neoplasia, with:
* No histological evidence of cancer with clinical follow-up data for a period of at least five years; or
* OSCC development (histologic or documented evidence of invasive cancer).
* Patients who had archived biopsy tissue blocks of a previous oral lesion(s) meeting the above criteria and retained at the same clinical center.

Exclusion Criteria:

* Patients with oral lesions or dysplasia with no indication of OSCC development or follow-up data of less than five years in non-OSCC patients.
* Patients diagnosed with oral epithelial dysplasia concomitant with OSCC at the time of the biopsy's original pathology report or a subsequent clinical note of cancer progression within three months post-biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population are patients presenting with an OPMD who have received a biopsy of their lesion. The study sample will be composed of patients with previously biopsied OPMDs from contracted clinics.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 5 years
  Standard measures of accuracy calculated using cross-tabulation of predicted risk category and confirmed cancer progression over a 5-year period from biopsy
Survival analysis | 5 years
  Kaplan-Meier analyses to compare time to a positive diagnosis of oral cancer between patients/biopsies with a STRATICYTE™ classification of Low- and Elevated-Risk.

SECONDARY OUTCOMES:
AUC | 5 years
  Area under the receiver operator curve
C-index (Harrell's) | 5 years
  From all possible pairs of patients, compute the number of concordant and discordant pairs. Compute C-index as the proportion of all possible pairs that are concordant.

CONTACTS AND LOCATIONS:
Overall Officials: Simon W Young, DDS, MD, PhD, Principal Investigator — UTHealthHouston
Locations (5):
- United States (5):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Loma Linda University, Loma Linda, California
  - Minnesota Oral and Facial Surgery, Minneapolis, Minnesota
  - MD Anderson Cancer Cetner, Houston, Texas
  - UTHealth Houston School of Dentistry, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwang JTK, Dammling C, McCord C, McGuire T, Park EP, Filkowski J, Shaw E, McMullen S, Nwigwe A, Ekwaru JP, McGaw WT, Lung KE, Seikaly H, Renick B, Lin DM, Morlandt A, Pritzker KH, Darling MR. External Validation of Straticyte, a Quantitative Biomarker-Based Risk Assay in Predicting Oral Cancer. J Maxillofac Oral Surg. 2025 Oct;24(5):1351-1357. doi: 10.1007/s12663-024-02362-7. Epub 2024 Oct 29. PMID 41054469
- [Background] Ralhan R, Desouza LV, Matta A, Tripathi SC, Ghanny S, Datta Gupta S, Bahadur S, Siu KW. Discovery and verification of head-and-neck cancer biomarkers by differential protein expression analysis using iTRAQ labeling, multidimensional liquid chromatography, and tandem mass spectrometry. Mol Cell Proteomics. 2008 Jun;7(6):1162-73. doi: 10.1074/mcp.M700500-MCP200. Epub 2008 Mar 13. PMID 18339795
- [Background] Ralhan R, Desouza LV, Matta A, Tripathi SC, Ghanny S, Dattagupta S, Thakar A, Chauhan SS, Siu KW. iTRAQ-multidimensional liquid chromatography and tandem mass spectrometry-based identification of potential biomarkers of oral epithelial dysplasia and novel networks between inflammation and premalignancy. J Proteome Res. 2009 Jan;8(1):300-9. doi: 10.1021/pr800501j. PMID 19072117
- [Background] Tripathi SC, Matta A, Kaur J, Grigull J, Chauhan SS, Thakar A, Shukla NK, Duggal R, DattaGupta S, Ralhan R, Siu KW. Nuclear S100A7 is associated with poor prognosis in head and neck cancer. PLoS One. 2010 Aug 3;5(8):e11939. doi: 10.1371/journal.pone.0011939. PMID 20689826
- [Background] Kaur J, Matta A, Kak I, Srivastava G, Assi J, Leong I, Witterick I, Colgan TJ, Macmillan C, Siu KW, Walfish PG, Ralhan R. S100A7 overexpression is a predictive marker for high risk of malignant transformation in oral dysplasia. Int J Cancer. 2014 Mar 15;134(6):1379-88. doi: 10.1002/ijc.28473. Epub 2013 Oct 8. PMID 24122701
- [Background] Hwang JT, Gu YR, Shen M, Ralhan R, Walfish PG, Pritzker KP, Mock D. Individualized five-year risk assessment for oral premalignant lesion progression to cancer. Oral Surg Oral Med Oral Pathol Oral Radiol. 2017 Mar;123(3):374-381. doi: 10.1016/j.oooo.2016.11.004. Epub 2016 Nov 22. PMID 28110942
- See also: Medlior Health Outcomes Research — https://www.medlior.com/
- See also: Oral Cancer Foundation — https://oralcancerfoundation.org/
- See also: Proteocyte Diagnostics Inc. — https://proteocyte.com